CLINICAL TRIAL: NCT07193147
Title: A Single Dose Pharmacokinetic and Safety Study of GZR4 Injection in Subjects With Mild, Moderate, and Severe Hepatic Impairment and Normal Hepatic Function
Brief Title: Pharmacokinetic and Safety Study of GZR4 Injection in Subjects With Hepatic Impairment
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZR4-T2D-105
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Diabetes
Keywords: GZR4 insulin
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GZR4 injection (Experimental)
  Interventions: Drug: GZR4

INTERVENTIONS:
Drug: GZR4 — GZR4 s.c., single-dose

SUMMARY:
This is a multicenter, single-dose, open-label, parallel Phase 1 clinical study to evaluate the PK profile, safety, and tolerability of GZR4 Injection in subjects with mild, moderate, and severe hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be included in the study.

  1. Subjects must fully understand the study contents, study procedures and possible risks and voluntarily sign the informed consent form;
  2. Male or female subjects aged ≥ 18 years and ≤ 75 years;
  3. Subjects should have no plans for fertility, sperm, or egg donation during the study and for 8 weeks postdose. They should be willing to use effective contraceptive measures during the study and for 8 weeks postdose, be surgically sterilized, or be female subjects who have reached menopause.
  4. Only for Subjects with Hepatic Impairment: Subjects with chronic hepatic impairment caused by viral hepatitis, alcoholic liver disease, autoimmune hepatitis, or other reasons;
  5. Only for Subjects with Hepatic Impairment: Subjects with a prior diagnosis of hepatic cirrhosis confirmed through liver biopsy or other medical imaging techniques;
  6. Only for Subjects with Hepatic Impairment: Subjects who have not received albumin within 14 days and are classified as Class A, B, or C according to the Child-Pugh score, with hepatic impairment resulting from prior primary liver disorders;
  7. Only for Subjects with Hepatic Impairment: Subjects with normal or abnormal and not clinically significant vital signs, physical examination, laboratory tests (hematology, blood chemistry, coagulation function and urinalysis), 12-lead ECG, chest X-ray and B-ultrasonography.

Exclusion Criteria:

* Subjects who meet any of the following criteria should not be enrolled in this study.

  1. Subjects with an allergic constitution, including a history of severe drug allergy or drug allergic reactions, who are known to be allergic to the investigational drug or its excipients (glycerol, phenol, m-cresol, zinc acetate dihydrate, sodium chloride, and citric acid monohydrate);
  2. Subjects with decompensated cardiac failure (NYHA Class III or IV) or those diagnosed with or highly suspected of having unstable angina pectoris or acute myocardial infarction, as well as those with malignant arrhythmias (such as ventricular fibrillation and sustained ventricular tachycardia) within 3 months before screening; subjects with a history of heart valve replacement surgery, coronary artery bypass grafting, or other invasive cardiovascular procedures, including percutaneous coronary intervention, as well as those who have experienced ischemic or hemorrhagic strokes (excluding lacunar infarctions) or transient ischemic attacks within 6 months before screening;
  3. Subjects with any clinically symptomatic bacterial, viral, parasitic, or fungal infection requiring systemic anti-infective therapy at screening (excluding hepatitis B and C in the hepatic impairment group), those with a history of severe active infection within 1 month before screening, or those who developed any acute infection requiring systemic anti-infective therapy within 2 weeks predose;
  4. Subjects with a history of drug abuse or drug addiction within 1 year before screening. Additionally, subjects with a positive urine drug abuse screening result predose (that cannot be attributed to concomitant medication) or a positive alcohol screening result;
  5. Subjects who are heavy smokers or alcohol consumers within 6 months before screening (consuming ≥ 14 units of alcohol per week: 1 unit ≈ 360 mL of beer, 45 mL of spirits, or 150 mL of wine; smoking ≥ 5 cigarettes per day), or those unable to abstain from smoking and alcohol for 48 h predose and during the study;
  6. Subjects who ingest grapefruit juice, food or beverage rich in methylxanthine (such as coffee, tea, cola, chocolate and functional drinks) within 7 days prior to dosing, or have strenuous exercise and other factors affecting drug absorption, distribution, metabolism and excretion, and cannot withdraw during the study;
  7. Pregnant or lactating women, women of child-bearing potential (WOCBP) with positive pregnancy test results at screening, or female subjects who have engaged in unprotected sexual intercourse within 2 weeks before screening;
  8. Subjects who are unwilling or unable to comply with the study procedures specified in the protocol, or who are deemed unsuitable for participating in this clinical study by any investigator.
  9. Subjects with hepatic impairment ：Subjects with a history of chronic or serious diseases in the circulatory system, digestive system, urinary system, immune system, blood system, endocrine and metabolic system, or mental and nervous system, or those who have the above conditions at screening that may interfere with the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-11-04 (Estimated)

PRIMARY OUTCOMES:
Cmax | through study completion, an average of 29 days
  Maximum plasma concentration
AUC0-last | through study completion, an average of 29 days
  Area under the plasma concentration-time curve at 0 h to last observation time-point after a single dose.

SECONDARY OUTCOMES:
AUC0-inf | through study completion, an average of 29 days
  Area under the plasma concentration-time curve at 0 h to infinity after a single dose.
AUC0-168h | Through study completion, an average of 29 days
  Area under the plasma concentration-time curve from time zero to 168 hours
Tmax | Through study completion, an average of 29 days
  Time of Maximum Drug ConcentrationTime to Maximum aentration
TEAE | through study completion, an average of 29 days
  Treatment Emergent Adverse Event

CONTACTS AND LOCATIONS:
Locations (1):
- Gan & Lee Pharmaceuticals Shandong Co., Ltd., Linyi, Shandong, China